CLINICAL TRIAL: NCT01280968
Title: Improving the Efficacy of Anti-Nicotine Immunotherapy
Acronym: PETNic002
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexey Mukhin (Other)
Collaborators: Wake Forest University Health Sciences (Other); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Alexey Mukhin, Professor of Psychiatry and Behavioral Science, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Pro00019787
Record Dates: First submitted 2010-11-16; First posted 2011-01-21 (Estimated); Results first posted 2013-12-18 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-01

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Aluminum Hydroxide; aluminum sulfate; nicotine Qbeta vaccine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NIC002 Vaccine in Aluminum hydroxide (Experimental): 4 subcutaneous vaccinations were performed over the course of 3 months, with 4 weeks between each vaccination. The administered volume of 0.65 mL of sterile water contained 100 μg of NIC002 and 0.46 mg aluminum hydroxide.
  Interventions: Biological: NIC002 in Aluminum hydroxide (Alum)
- Placebo Vaccine - Aluminum hydroxide (Placebo Comparator): 4 placebo injections were administered subcutaneously over the course of 3 months, with 4 weeks between each vaccination. The administered volume of 0.65 mL of sterile water contained 0.46 mg aluminum hydroxide.
  Interventions: Biological: Placebo Vaccine - Aluminum hydroxide

INTERVENTIONS:
Biological: NIC002 in Aluminum hydroxide (Alum) — Fifty-five subjects will receive 4 subcutaneous injections of 0.1 mg Nicotine-QB (NIC002) in Alum vaccine with a 4-week interval between injections.
  Other Names: CYT002-NicQb (Nicotine-Qbeta); Anti-Nicotine Vaccine
  Arms: NIC002 Vaccine in Aluminum hydroxide
Biological: Placebo Vaccine - Aluminum hydroxide — Ten subjects will receive 4 subcutaneous injections of indistinguishable placebo (Alum alone) with a 4-week interval between injections.
  Arms: Placebo Vaccine - Aluminum hydroxide

SUMMARY:
The purpose of this study is to find out how vaccine-induced antibodies change the way the body processes nicotine from cigarettes. These antibodies absorb nicotine and can reduce nicotine levels in the brain. In this way, the vaccination may help to quit smoking. The central hypothesis is that anti-nicotine antibodies change kinetics of brain nicotine accumulation and distribution of nicotine between the brain and other body tissues. This vaccine is investigational which means that it is still being tested in research studies and is not approved by the U.S. Food and Drug Administration (FDA) to help people quit smoking.

ELIGIBILITY:
Inclusion Criteria:

* 18-55 years old
* Smoked an average of at least 10 cigarettes per day for the past year
* Have an expired air Carbon Monoxide (CO) reading of at least 15 ppm
* Express a desire to quit smoking in the next three to four months.
* Potential subjects must agree to use acceptable contraception during their participation in this study.
* Potential subjects must agree to avoid the following during their participation in this study:
* participation in any other nicotine-related modification strategy outside of this protocol
* use of tobacco products other than cigarettes, including pipe tobacco, cigars, snuff, and chewing tobacco

  * use of experimental (investigational) drugs or devices;
  * use of illegal drugs;
  * use of psychiatric medications;
  * use of opiate medications;
  * use of systemic steroids or other immunosuppressive agents.

Exclusion Criteria:

1. Hypertension (systolic >140 mm Hg, diastolic >100 mm Hg, coupled with a history of hypertension); subjects with no previous diagnosis of hypertension may have a screening blood pressure up to 160/100.
2. Hypotension with symptoms (systolic <90 mm Hg, diastolic <60 mm Hg).
3. Participants with a history of hypertension may, however, be allowed to participate in the study if the study physician or physician assistant determines that the condition is stable, controlled by medication, and in no way jeopardizes the individual's safety.
4. Coronary heart disease or other cardiovascular disorder;
5. Lifetime history of heart attack;
6. Cardiac rhythm disorder (irregular heart rhythm);
7. Chest pains (unless history, exam, and Electrocardiogram (ECG) clearly indicate a non-cardiac source);
8. Cardiac (heart) disorder (including but not limited to valvular heart disease, heart murmur, heart failure);
9. Liver or kidney disorder (except kidney stones, gallstones);
10. Gastrointestinal problems or disease other than gastroesophageal reflux or heartburn;
11. Active ulcers in the past 30 days;
12. Lung disorder (including but not limited to chronic obstructive pulmonary disease (COPD), emphysema, and asthma);
13. Brain abnormality or other neurological disorder (including but not limited to stroke, brain tumor, and seizure disorder);
14. Recent, unexplained fainting spells;
15. Problems giving blood samples;
16. Diabetes treated with insulin; non-insulin treated diabetes (unless glucose is less than 180mg/dcl and HbA1c is less than 7%);
17. Current cancer or treatment for cancer in the past six months (except basal or squamous cell skin cancer);
18. Skin disorder;
19. Autoimmune disease;
20. Human immunodeficiency virus (HIV) or HIV risk behavior;
21. Severe allergies;
22. Other major medical condition;
23. Current psychiatric disease including major depressive episode, panic attack, psychosis, bipolar disorder or eating disorder;
24. Pregnant or nursing mothers;
25. Use (within the past 30 days) of:

    * Illegal drugs (or if the urine drug screen is positive),
    * Experimental (investigational) drugs;
    * Psychiatric medications including antidepressants, anti-psychotics or any other medications that are known to affect smoking cessation (e.g. clonidine);
    * Opiate medications for pain or sleep (non-opiate medication for pain or sleep will be allowed)
    * Smokeless tobacco (chewing tobacco, snuff), cigars, pipes or e-cigarettes;
    * Nicotine replacement therapy or any other smoking cessation aid.
26. Alcohol abuse - The AUDIT (Alcohol Use Disorders Identification Test) questionnaire will be used to assess alcohol abuse.
27. Previous history of negative experiences with "flu" vaccine or any other vaccine.
28. High chronic exposure to aluminum (occupational or medical);
29. Pulmonary function test results < 60% of predicted value for FEV1 and FVC;
30. Body Mass Index > 38kg/m2;
31. History of psychosis or bipolar disorder;
32. Prior exposure to CTY002- NicQ or any other nicotine vaccine.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2010-12; Primary Completion 2012-09 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexey G Mukhin, M.D., Ph.D., Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke Center for Nicotine & Smoking Cessation Research, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NIC002 Vaccine in Aluminum Hydroxide | Placebo Vaccine - Aluminum Hydroxide
Started | 45 | 7
Completed | 27 | 4
Not Completed | 18 | 3
Not completed — Lost to Follow-up | 8 | 2
Not completed — Unable to Follow Experimental Protocol | 2 | 0
Not completed — Commuting Problems | 2 | 0
Not completed — Anxiety | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Scheduling Conflicts | 1 | 1
Not completed — Pre-existing Neurological Condition | 1 | 0
Not completed — Unable to Smoke in Supine Position | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NIC002 Vaccine in Aluminum Hydroxide | Placebo Vaccine - Aluminum Hydroxide | Total
Number analyzed (Participants) | 45 | 7 | 52
Age, Customized [Mean (Full Range); unit: years] — One participant reported that she was 54 at the screening, but after she was consented, it was discovered that she was actually 56. However, the subject was discontinued after the first study visit because she could not use the smoking delivery device; therefore, she received no vaccinations. Safety Event #14 was submitted to Duke IRB to account for this Protocol Deviation in which the subject was out of the age range.
  years | 43 [23 to 56] | 44 [35 to 55] | 43 [23 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 4 | 26
  Male | 23 | 3 | 26
Region of Enrollment [Number; unit: participants]
  United States | 45 | 7 | 52
Cigarettes Per Day [Mean (Full Range); unit: cigarettes per day] — average number of cigarettes participant smokes each day
  cigarettes per day | 19 [10 to 30] | 21 [16 to 30] | 19 [10 to 30]
Pack-Years [Mean (Full Range); unit: pack-years] — pack-years that each participant has smoked, calculated by multiplying the number of packs of cigarettes participant smokes each day by number of years participant has smoked
  pack-years | 22 [4 to 45] | 25 [18 to 32] | 22 [4 to 45]

OUTCOME MEASURES:

1. Primary Outcome: Vaccine-Induced Percent Change in Brain Nicotine Area Under Curve (AUC) After Single or Multiple (7) Puffs
Description: There was a 2 hour washout period between the "single puff" and "multiple puffs" assessments.
Time Frame: measured at week 1 and week 16
Measure: Mean (Standard Error); unit: percentage of change
Groups:
- NIC002 Vaccine in Aluminum Hydroxide, All Vaccinated Subjects: 4 subcutaneous vaccinations were performed over the course of 3 months, with 4 weeks between each vaccination. The administered volume of 0.65 mL of sterile water contained 100 μg of NIC002 and 0.46 mg aluminum hydroxide.
Arm/Group | NIC002 Vaccine in Aluminum Hydroxide, All Vaccinated Subjects | NIC002, Tertile With Highest Antibody Binding Capacity | Placebo Vaccine - Aluminum Hydroxide
Number analyzed (Participants) | 29 | 10 | 4
percentage of change
  single cigarette puff | 1 (5) | -15 (7) | -0.2 (7.1)
  multiple cigarette puffs | 0.1 (5.7) | -9 (8) | -1.1 (9.6)

2. Primary Outcome: Vaccine-Induced Percent Change in Brain Nicotine Maximum Concentration After Single or Multiple (7) Puffs
Description: There was a 2 hour washout period between the "single puff" and "multiple puffs" assessments.
Time Frame: measured at week 1 and week 16
Measure: Mean (Standard Error); unit: percentage of change
Arm/Group | NIC002 Vaccine in Aluminum Hydroxide, All Vaccinated Subjects | NIC002, Tertile With Highest Antibody Binding Capacity | Placebo Vaccine - Aluminum Hydroxide
Number analyzed (Participants) | 29 | 10 | 4
percentage of change
  single cigarette puff | 1 (4) | -15 (6) | 0 (7.8)
  multiple cigarette puffs | -0.7 (5.1) | -6 (9) | -1.3 (9.8)

3. Primary Outcome: Vaccination-Induced Percent Change in T1/2 of Brain Nicotine Accumulation After Single or Multiple (7) Puffs
Description: There was a 2 hour washout period between the "single puff" and "multiple puffs" assessments.
Time Frame: measured at week 1 and week 16
Measure: Mean (Standard Error); unit: percentage of change
Arm/Group | NIC002 Vaccine in Aluminum Hydroxide, All Vaccinated Subjects | NIC002, Tertile With Highest Antibody Binding Capacity | Placebo Vaccine - Aluminum Hydroxide
Number analyzed (Participants) | 29 | 10 | 4
percentage of change
  single cigarette puff | 0 (11) | 15 (30) | -4.4 (9.6)
  multiple cigarette puffs | -2 (4) | 0 (7) | 3.8 (11.6)

4. Primary Outcome: Vaccination-Induced Percent Change in Initial Slope of Brain Nicotine Accumulation After a Single Puff
Time Frame: measured at week 1 and week 16
Measure: Mean (Standard Error); unit: percentage of change
Arm/Group | NIC002 Vaccine in Aluminum Hydroxide, All Vaccinated Subjects | NIC002, Tertile With Highest Antibody Binding Capacity | Placebo Vaccine - Aluminum Hydroxide
Number analyzed (Participants) | 29 | 10 | 4
percentage of change | 22.5 (12.7) | 9 (30) | 2.4 (5.9)

ADVERSE EVENTS:
Description: The number of participants at risk is different from the number of enrolled participants because not all participants who were randomized to a vaccine or placebo received treatment. Of the 52 participants who were assigned to a treatment group, only 41 received at least one vaccination. Therefore, 41 participants were at risk.
Arm/Group | NIC002 Vaccine in Aluminum Hydroxide | Placebo Vaccine - Aluminum Hydroxide
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/5
Other Adverse Events (participants affected / at risk) | 13/36 | 3/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NIC002 Vaccine in Aluminum Hydroxide (N=36) | Placebo Vaccine - Aluminum Hydroxide (N=5)
Headache (General disorders) | 3 (8) | 1 (1) — At each of 8 visits following first vaccination visit, participants filled out Side Effects Questionnaire and rated severity of side effect from 1 (not at all) to 7 (extremely). Adverse events represent side effects rated as 5 (a lot) or higher.
Weight Changes (General disorders) | 1 (2) | 1 (1) — At each of 8 visits following first vaccination visit, participants filled out Side Effects Questionnaire and rated severity of side effect from 1 (not at all) to 7 (extremely). Adverse events represent side effects rated as 5 (a lot) or higher.
Back Pain (General disorders) | 2 (2) | 0 (0) — At each of 8 visits following first vaccination visit, participants filled out Side Effects Questionnaire and rated severity of side effect from 1 (not at all) to 7 (extremely). Adverse events represent side effects rated as 5 (a lot) or higher.
Feeling Cold (General disorders) | 3 (9) | 0 (0) — At each of 8 visits following first vaccination visit, participants filled out Side Effects Questionnaire and rated severity of side effect from 1 (not at all) to 7 (extremely). Adverse events represent side effects rated as 5 (a lot) or higher.
Feeling Hot (General disorders) | 4 (5) | 0 (0) — At each of 8 visits following first vaccination visit, participants filled out Side Effects Questionnaire and rated severity of side effect from 1 (not at all) to 7 (extremely). Adverse events represent side effects rated as 5 (a lot) or higher.
Nasal Congestion (General disorders) | 0 (0) | 1 (1) — At each of 8 visits following first vaccination visit, participants filled out Side Effects Questionnaire and rated severity of side effect from 1 (not at all) to 7 (extremely). Adverse events represent side effects rated as 5 (a lot) or higher.
Runny Nose (General disorders) | 0 (0) | 1 (1) — At each of 8 visits following first vaccination visit, participants filled out Side Effects Questionnaire and rated severity of side effect from 1 (not at all) to 7 (extremely). Adverse events represent side effects rated as 5 (a lot) or higher.
Sore Throat (General disorders) | 2 (2) | 0 (0) — At each of 8 visits following first vaccination visit, participants filled out Side Effects Questionnaire and rated severity of side effect from 1 (not at all) to 7 (extremely). Adverse events represent side effects rated as 5 (a lot) or higher.
Fatigue (General disorders) | 4 (11) | 1 (1) — At each of 8 visits following first vaccination visit, participants filled out Side Effects Questionnaire and rated severity of side effect from 1 (not at all) to 7 (extremely). Adverse events represent side effects rated as 5 (a lot) or higher.
Tenderness at Injection Site (General disorders) | 2 (2) | 0 (0) — At each of 8 visits following first vaccination visit, participants filled out Side Effects Questionnaire and rated severity of side effect from 1 (not at all) to 7 (extremely). Adverse events represent side effects rated as 5 (a lot) or higher.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No